CLINICAL TRIAL: NCT00053443
Title: Compliance Enhancement In HIV/AIDS Patients
Brief Title: Handheld Computers to Improve Adherence to Anti-HIV Drug Regimens
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: 2R44AI43750-02 A 2; 5R44AI043750-03 (NIH)
Record Dates: First submitted 2003-01-29; First posted 2003-01-30 (Estimated); Last update posted 2016-12-14 (Estimated); Status verified 2005-12

CONDITIONS: HIV Infections
Keywords: Adherence; Treatment Experienced
MeSH Terms: conditions — HIV Infections

INTERVENTIONS:
Device: Medication Reminder System/Adherence Tracker

SUMMARY:
While anti-HIV drugs can significantly reduce viral loads, the medication regimens can be complex, and patients must take them correctly for the best effect. Nonadherent patients risk developing drug resistant HIV strains. The purpose of this study is to evaluate the effectiveness of a handheld computerized system designed to help patients take their drugs correctly.

DETAILED DESCRIPTION:
As the use of protease inhibitors and other antiretroviral medications has increased, multiple drug resistant HIV strains have emerged, demonstrating the need for improved patient adherence to complex drug regimens. Individual computerized adherence systems have been proposed as a mechanism for improving patient adherence. This study will utilize advanced computer and communication technologies to produce a handheld (PDA) product for HIV/AIDS patients. The system serves as a patient reminder system, addresses problems of missed medications, and monitors severity of side effects. This study will evaluate the efficacy of the system as an adherence intervention.

Participants in the study will be randomized to either the intervention or a control group. Participants will use the PDA daily for medication reminders, alarms, adherence tracking, and as a source of information on HIV/AIDS. The study will last 15 weeks. Each participant will have 6 study interviews and 2 quality control interviews. Study interviews will include adherence questionnaires, blood tests for viral load and CD4 data, and quality of life assessments.

ELIGIBILITY:
Inclusion Criteria

* HIV positive
* Currently taking medications for HIV/AIDS.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 156
Dates: Primary Completion 2005-12 (Actual); Study Completion 2005-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Inflexxion, Newton, Massachusetts, United States